CLINICAL TRIAL: NCT06307886
Title: Comparison of Five-year Survival and Disease-free Survival in Patients Diagnosed With Endometrium Cancer Who Underwent Total Laparoscopic Hysterectomy With and Without Uterine Manipulator
Status: Recruiting | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: GaziosmanpasaTREHSs
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients diagnosed with endometrium cancer
  Interventions: Procedure: Patients Diagnosed With Endometrium Cancer Who Underwent Total Laparoscopic Hysterectomy With manipulator; Procedure: lPatients Diagnosed With Endometrium Cancer Who Underwent Total Laparoscopic Hysterectomy without uterine manipulator

INTERVENTIONS:
Procedure: Patients Diagnosed With Endometrium Cancer Who Underwent Total Laparoscopic Hysterectomy With manipulator — patients who underwent laparoscopic hysterectomy with using uterine manipulator
Procedure: lPatients Diagnosed With Endometrium Cancer Who Underwent Total Laparoscopic Hysterectomy without uterine manipulator — patients who underwent laparoscopic hysterectomy without using uterine manipulator

SUMMARY:
Comparison of five-year survival and disease-free survival in patients diagnosed with endometrium cancer who underwent total laparoscopic hysterectomy with and without a uterine manipulator

ELIGIBILITY:
Inclusion Criteria:

* patients suitable for laparoscopic surgery patients ages 18-75 patients diagnosed figo stage 1 and 2 endometrial cancer

Exclusion Criteria:

* patients not suitable for laparoscopic surgery patients diagnosed figo stage 3 and 4 endometrial cancer pregnant patients

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients Diagnosed With Endometrium Cancer Who Underwent Total Laparoscopic Hysterectomy With and Without Uterine Manipulator
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
five year survival in patients diagnosed with endometrial cancer | 5 year
disease-free survival in patients diagnosed with endometrial cancer | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Training and research hospital, Istanbul, Turkey (Türkiye)